CLINICAL TRIAL: NCT01824745
Title: Survivorship Care Planning for At Risk Breast Cancer Survivors
Brief Title: Survivorship Care Planning in Improving the Quality of Life in Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12383; NCI-2013-00734 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Cancer Survivor
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Methods; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (SCP-BCS template booklet and counseling) (Experimental): Participants receive SCP-BCS template booklet and receive counseling sessions with a patient navigator for 40 minutes twice weekly for 4 sessions.
  Interventions: Other: educational intervention; Other: counseling intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm II (SCP-BCS template booklet) (Active Comparator): Participants receive SCP-BCS template booklet and receive standard follow-up care.
  Interventions: Other: educational intervention; Procedure: standard follow-up care; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Other: educational intervention — Receive the SCP-BCS template booklet
  Other Names: intervention, educational
Other: counseling intervention — Receive counseling sessions with a patient navigator
  Other Names: counseling and communications studies
  Arms: Arm I (SCP-BCS template booklet and counseling)
Procedure: standard follow-up care — Receive standard follow-up care
  Arms: Arm II (SCP-BCS template booklet)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies survivorship care planning in improving the quality of life in breast cancer survivors. Survivorship care planning may reduce stress and improve the well-being and quality of life of cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the effectiveness of the navigation intervention and survivorship care plan (SCP)-breast cancer survivors (BCS) template booklet on accessing and adhering to SCP-BCS guidelines compared to the control group receiving usual care and the SCP-BCS template booklet.

SECONDARY OBJECTIVES:

I. Develop a clinically and psychosocially responsive SCP-breast cancer survivors (SCP-BCS) template in English and English-Spanish adopted from American Society of Clinical Oncology (ASCO)-SCP.

II. Assess the acceptability, utility and format preference (electronic vs paper) of the SCP-BCS template.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive SCP-BCS template booklet and receive counseling sessions with a patient navigator for 40 minutes twice weekly for 4 sessions.

ARM II: Participants receive SCP-BCS template booklet and receive standard follow-up care.

After completion so study treatment, participants are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* In early survivorship phase, defined as being post-surgery to ending of active treatment to 18 months post active treatment for stage 0-3 breast cancer (BCA)
* Reside in Southern California
* BCS treated at Kaiser, an health maintenance organization (HMO) provider, will be excluded since their SCP implementation project is underway
* BCS will not be excluded based on cancer treatments received or a history of diagnosis of mild depression, anxiety, and hypertension and diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07-15; Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of BCS accessing a SCP from their oncology provider | At 6 months
  Fisher's exact test will be used to test the null hypothesis (at least 40% of trial participants will have access to SCP).

SECONDARY OUTCOMES:
Adherence to SCP guidelines | At 12 months
  Fisher's exact test will be used to test the null hypothesis (at least 25% of participants reporting adherence to SCP guidelines).
Proportion of BCS accessing a SCP from their oncology provider | At 12 months
  Fisher's exact test will be used to test the null hypothesis (at least 60% of trial participants will have access to SCP).

OTHER OUTCOMES:
Develop a clinically and psychosocially responsive SCP-BCS template in English and a linguistically response bilingual version (English-Spanish) | Up to 12 months
  The acceptability, utility, and format preference will also be assessed. A rating score will be generated for acceptability and utility and 95% confidence intervals for the proportion of BCS rating score at >= 4 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kimlin Ashing-Giwa, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California